CLINICAL TRIAL: NCT03367234
Title: A Simple Large Trial of Patient-Centered Care for Opioid Use Disorders in Federally Qualified Healthcare Centers and Specialty Care Settings
Brief Title: Patient-Centered Care for Opioid Use Disorders in Federally Qualified Healthcare Centers and Specialty Care Settings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study experienced delays due to site recruitment. Funder terminated contract.
Sponsor: Public Health Management Corporation (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS-1605-35373
Record Dates: First submitted 2017-11-28; First posted 2017-12-08 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Opioid-use Disorder; Substance Use Disorders
Keywords: Federally Qualified Health Center; Contingency Management; Cognitive Behavioral Therapy; Cognitive Behavioral / Relapse Prevention; Medication Assisted Treatment; Behavioral Health Consultant; Integrated Care
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy; Opiate Substitution Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Addiction-to-Health (PATH) (Experimental): Cognitive Behavioral Therapy (CBT) sessions with a behavioral health consultant twice weekly for weeks 1-13, once weekly for weeks 14-26, as needed weeks 27-52; Contingency management rewards for specified recovery behaviors which could include medication adherence, attendance at CB/RP sessions and/or CB/RP exercise participation; Medication-assisted treatment, either extended-release naltrexone once monthly or buprenorphine once daily; Peer recovery specialist support twice weekly for weeks 1-13, once weekly for weeks 14-26, as needed for weeks 27-52; Psychiatric consultation as needed.
  Interventions: Behavioral: Individual Therapy Sessions; Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Medication-Assisted Treatment; Behavioral: Peer Recovery Specialist Support; Behavioral: Psychiatric Consultation; Behavioral: Contingency Management
- Standard Care (Active Comparator): Treatment may differ slightly by treatment program, but addiction specialty Intensive Outpatient Treatment (ASAM Level 2.1) will generally include individual therapy sessions with a counselor 1 hour per week for week; Medication-assisted treatment, either extended-release naltrexone once monthly or suboxone once daily; Group therapy sessions 9 hours per week then decreasing to 3 hours per week; Psychiatric consultation as needed.
  Interventions: Behavioral: Individual Therapy Sessions; Behavioral: Medication-Assisted Treatment; Behavioral: Peer Recovery Specialist Support; Behavioral: Group Therapy Sessions; Behavioral: Psychiatric Consultation

INTERVENTIONS:
Behavioral: Individual Therapy Sessions — One-on-one sessions with a counselor
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive Behavioral Therapy techniques delivered by a behavioral health consultant (BHC)
  Other Names: CBT; CB/RP
  Arms: Personalized Addiction-to-Health (PATH)
Behavioral: Medication-Assisted Treatment — Buprenorphine or Extended-Release Naltrexone
  Other Names: MAT
Behavioral: Peer Recovery Specialist Support — Individual and/or group sessions with a certified peer recovery specialist
Behavioral: Group Therapy Sessions — Group therapy sessions
  Arms: Standard Care
Behavioral: Psychiatric Consultation — Access to psychiatric consultation
Behavioral: Contingency Management — Rewards for engagement in specified recovery behaviors
  Arms: Personalized Addiction-to-Health (PATH)

SUMMARY:
This study evaluates the effectiveness of integrating empirically-supported treatments for an opioid use disorder into a primary care setting. These treatments will include ASAM Criteria multidimensional assessment, cognitive behavioral therapy and relapse prevention with contingency management, medication-assisted treatment, and recovery support services. Half of participants will be assigned to opioid use disorder treatment in a federally qualified health center, and half will receive treatment at a publicly-funded intensive outpatient addiction treatment program which has the ability to offer medication-assisted treatment.

DETAILED DESCRIPTION:
This is a large, simple, comparative effectiveness trial of the Personalized Addiction Treatment-to-Health Model vs. standard care in the community specialty addiction treatment system. PATH combines several empirically supported treatment methods in a flexible schedule in tandem with primary care, with the goals of higher rates of confirmed substance abstinence and treatment retention.

PATH components include: 1) The CONTINUUM multidimensional assessment, an evidence-based implementation of the American Society of Addiction Medicine (ASAM) placement criteria; 2) Cognitive Behavioral Relapse Prevention (CB/RP), a skills-based approach centered on teaching coping skills to handle risky situations that can be practiced and learned; 3) Contingency management (CM), which targets chronic substance use's diminution of brain dopaminergic reward by specifically conditioning positive recovery behaviors via immediate financial incentives; and 4) Recovery Support Services, non-professional community-based services for wrap-around care needs.

Effect sizes for a combined CB/RP and CM approach appear to be large and there is evidence that this combination results in longer lasting improvements presumably as homeostasis returns to the reward system. An extensive literature demonstrates that counseling plus medication-assisted treatment (MAT) yields superior outcomes versus counseling alone. Buprenorphine and extended-release naltrexone are well suited for use in primary care. Buprenorphine is a partial agonist at the mu-opioid receptor that provides anti-withdrawal and anti-craving effects for up to 36 hours on a single dose. Partial agonism and a slow onset diminish the patient's perception of euphoria, limiting abuse, while the long half-life and binding duration make it useful for both detoxification and long-term opioid maintenance. Extended-release naltrexone is a once-monthly intramuscular injection that, following detoxification, provides opioid receptor blockade for at least 30 days and is safe and effective for prolonging abstinence and preventing relapse from opiates.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years or older
2. As determined according to the ASAM Criteria CONTINUUM Software decision engine, patient meets criteria for: a) Level 1 care, i.e., outpatient treatment, OR b) Level 2 care, i.e., intensive outpatient treatment.

Exclusion Criteria:

1. The medical practitioner or BHC overrule these criteria because medical and psychiatric complications exist that would contraindicate research participation
2. Patient requires an ASAM level of care greater than Level 2
3. The patient reports plans to leave the area (i.e. Philadelphia or Washington, DC greater metropolitan area) within the next 6 months
4. The patient is not English-speaking
5. The patient is unable to provide valid informed consent by correctly describing the key components of consent to the Research Assistant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in confirmed substance abstinence | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  On-site urine drug testing kits rapidly test for cocaine, opiates, amphetamines, methamphetamines, benzodiazepines, cannabis, barbiturates, Phencyclidine, and alcohol. Urine testing will be administered at all follow-ups to capture use within the last 3 days.
Change in retention in treatment | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  Verify patient self-report of treatment engagement by acquiring payment data from funders. Federally Qualified Health Centers and Standard Care Intensive Outpatient programs will release study patient records to resolve inconsistencies between patient report and billing data, including treatment session attendance, medications prescribed, prescriptions filled, doses received, and results from urinalysis testing. Data will be collected for the past 3 months.

SECONDARY OUTCOMES:
Lower rates of service utilization | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  Patient reported service utilization including substance abuse treatment, medical services, visits to medical offices, hospitalizations, and emergency room visits received that were not a part of the assigned treatment during the past 3 months
Higher quality of life | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  Self-reported enjoyment and satisfaction experienced in various areas of daily functioning during the past week
Lower rates of HIV risk behaviors | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  Self-reported drug use, injection-related risk behavior, sexual risk, and HIV testing history and results for the past 3 months.

OTHER OUTCOMES:
Change in Employment Severity Score | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  The American Society of Addiction Medicine (ASAM) Continuum is computer-guided, standardized interview for assessing and caring for patients with substance use disorders and co-occurring conditions. The employment section asks participants about their employment status during the past 3 months using questions from the Addiction Severity Index (ASI). The composite score of the ASI employment section ranges from 0-1 with higher scores indicating greater problem severity.
Change in Family/Social Functioning Severity Score | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  The American Society of Addiction Medicine (ASAM) Continuum is computer-guided, standardized interview for assessing and caring for patients with substance use disorders and co-occurring conditions. The family and social functioning section asks participants about their family and social functioning during the past 3 months using questions from the Addiction Severity Index (ASI). The composite score of the ASI family and social functioning section ranges from 0-1 with higher scores indicating greater problem severity.
Change in Psychiatric Severity Score | Baseline, 3-, 6-, 9-, 12-, 15-, and 18 month follow-ups
  The American Society of Addiction Medicine (ASAM) Continuum is computer-guided, standardized interview for assessing and caring for patients with substance use disorders and co-occurring conditions. The psychiatric section asks participants about their psychiatric functioning during the past 3 months using questions from the Addiction Severity Index (ASI). The composite score of the ASI psychiatric section ranges from 0-1 with higher scores indicating greater problem severity.

CONTACTS AND LOCATIONS:
Overall Officials: David R Gastfriend, MD, Principal Investigator — Public Health Management Corporation

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03367234/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03367234/SAP_001.pdf